CLINICAL TRIAL: NCT04175990
Title: Role Of Dydrogesterone Towards Oocyte and Embryo Quality in Polycystic Ovarian Syndrome (PCOS)
Brief Title: IVF Outcome Following Progestogen Ovarian Stimulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azrai Abu, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UKMPPI/111/8/JEP-2018-165
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: IVF; Oocyte Maturation Defect 1; Clinical Pregnancy Rate; Ovarian Hyperstimulation
Keywords: progestogen; ovarian stimulation regime; IVF outcome
MeSH Terms: interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progestogen (Experimental): Oral Dydrogesterone 10mg tds was given from day 1 of menses till day of trigger
  Interventions: Drug: Dydrogesterone Pill
- standard combine minimal stimulation protocol (No Intervention): Oral clomiphene citrate 100mg daily given from day 1 till day 10 of menses with additional gonadotrophin (Menopur 225mg daily) from day 3 of menses till trigger day

INTERVENTIONS:
Drug: Dydrogesterone Pill — started from day 1 of menses till trigger day
  Arms: Progestogen

SUMMARY:
The new strategy is by using the progestogen to block the luteinizing hormone(LH) surge either endogenous during luteal phase stimulation, or exogenous in the follicular phase i.e progestin primed ovarian stimulation (PPOS). The goal of PPOS is to develop a single dominant follicle. Various types of oral Progestin had been studied before including Medroxyprogesterone Acetate (MPA) and Utrogestan with different dosage. A different study by Wang et al conducted by using MPA to patients with PCOS. The use of MPA is contraindicated in human pregnancy whereas Dydrogesterone had been extensively used worldwide for the treatment of threatened miscarriage as well as luteal support in infertility setting. Previous protocol on PPOS showed inconclusive results. Therefore in this study, Dydrogesterone was used as the Progestin Primed Ovarian hyperstimulation to explore its effect on PCOS women IVF outcome.

DETAILED DESCRIPTION:
This is a prospective controlled cohort study conducted at the Department of Medical Assisted Conception (MAC) unit of the University Kebangsaan Malaysia Medical Centre (UKMMC). From May 2018 through May 2019, women with Polycystic Ovarian Syndrome (PCOS) undergoing IVF/intracytoplasmic sperm insemination(ICSI) regimens for the treatment of infertility were recruited.

Patients recruited will then be randomized accordingly using the randomizer software. Group A will be the interventional group and group B will be the control group.

Oocyte retrieval will be performed 34-36 hours following the human chorionic gonadotrophin (hCG) trigger. Sperm was obtained on the same day. Mature oocytes will be fertilized with sperm via IVF or ICSI. Fertilized embryos were observed via time laps method and the progress and cleavage were monitored before planning for embryo transfer. Embryo transfer will be performed on day 3 or day 5 after oocyte retrieval.

All results will be analyzed using Statistical Package for the Social Sciences(SPSS) version 21 software. Descriptive analysis will be done for demographic data and presented in mean ± Standard deviation (SD). Demographic characteristic between the two groups will be compared with the use of the Mann-Whitney U test. The categorical data was analysed by using Chi-square test for the association of variables. A p-value of 0.05 or less was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

* · Aged 20 - 40 years old

  * Basal serum follicular stimulating hormone(FSH) level of no more than 10 IU/L
  * Diagnosis of PCOS met using Rotterdam criteria.

Exclusion Criteria:

* low AMH level (AMH less than 3 ng/ml).

  * Contraindicated to ovarian stimulation treatment eg: history of severe ovarian hyper stimulation syndrome(OHSS)
  * Presence of uterine pathology eg: adenomyosis, large uterine fibroid.
  * Patients who has had poor ovarian stimulation of twice or more.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Number of oocyte retrieval | 30 hour after trigger with HCG 10000 International unit (IU)
  number of oocyte retrieved
Biochemical pregnancy rate | 14 days after embryo transferred
  serum Bhcg more than 5 mol/L
clinical pregnancy rate | 4 weeks after embryo transfer
  presence of intrauterine gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad azrai abu, medical Degree, Principal Investigator — Department of Obstetrics and Gynecology, UKM Medical Centre
Locations (1):
- Medically Assisted Conception Unit, Ukm Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 7. Neill JD. Knobil and Neill's physiology of reproduction. 3rd edition. San Diego, CA: Elsevier, 2006: 1289-301
- [Result] Lizneva D, Suturina L, Walker W, Brakta S, Gavrilova-Jordan L, Azziz R. Criteria, prevalence, and phenotypes of polycystic ovary syndrome. Fertil Steril. 2016 Jul;106(1):6-15. doi: 10.1016/j.fertnstert.2016.05.003. Epub 2016 May 24. PMID 27233760
- [Result] Boomsma CM, Fauser BC, Macklon NS. Pregnancy complications in women with polycystic ovary syndrome. Semin Reprod Med. 2008 Jan;26(1):72-84. doi: 10.1055/s-2007-992927. PMID 18181085
- [Result] Sam S, Dunaif A. Polycystic ovary syndrome: syndrome XX? Trends Endocrinol Metab. 2003 Oct;14(8):365-70. doi: 10.1016/j.tem.2003.08.002. PMID 14516934
- [Result] Shah DK, Missmer SA, Berry KF, Racowsky C, Ginsburg ES. Effect of obesity on oocyte and embryo quality in women undergoing in vitro fertilization. Obstet Gynecol. 2011 Jul;118(1):63-70. doi: 10.1097/AOG.0b013e31821fd360. PMID 21691164
- [Result] Zhu X, Ye H, Fu Y. The Utrogestan and hMG protocol in patients with polycystic ovarian syndrome undergoing controlled ovarian hyperstimulation during IVF/ICSI treatments. Medicine (Baltimore). 2016 Jul;95(28):e4193. doi: 10.1097/MD.0000000000004193. PMID 27428219
- [Result] Al-Inany HG, Youssef MA, Ayeleke RO, Brown J, Lam WS, Broekmans FJ. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD001750. doi: 10.1002/14651858.CD001750.pub4. PMID 27126581
- [Result] van der Spuy ZM, Dyer SJ. The pathogenesis of infertility and early pregnancy loss in polycystic ovary syndrome. Best Pract Res Clin Obstet Gynaecol. 2004 Oct;18(5):755-71. doi: 10.1016/j.bpobgyn.2004.06.001. PMID 15380145
- [Result] Bosch E, Valencia I, Escudero E, Crespo J, Simon C, Remohi J, Pellicer A. Premature luteinization during gonadotropin-releasing hormone antagonist cycles and its relationship with in vitro fertilization outcome. Fertil Steril. 2003 Dec;80(6):1444-9. doi: 10.1016/j.fertnstert.2003.07.002. PMID 14667881
- [Result] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Result] Wang Y, Chen Q, Wang N, Chen H, Lyu Q, Kuang Y. Controlled Ovarian Stimulation Using Medroxyprogesterone Acetate and hMG in Patients With Polycystic Ovary Syndrome Treated for IVF: A Double-Blind Randomized Crossover Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2939. doi: 10.1097/MD.0000000000002939. PMID 26945402
- [Result] Zhu X, Zhang X, Fu Y. Utrogestan as an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Medicine (Baltimore). 2015 May;94(21):e909. doi: 10.1097/MD.0000000000000909. PMID 26020402
- [Result] McCartney CR, Marshall JC. CLINICAL PRACTICE. Polycystic Ovary Syndrome. N Engl J Med. 2016 Jul 7;375(1):54-64. doi: 10.1056/NEJMcp1514916. PMID 27406348
- [Result] Diamond MP, Kruger M, Santoro N, Zhang H, Casson P, Schlaff W, Coutifaris C, Brzyski R, Christman G, Carr BR, McGovern PG, Cataldo NA, Steinkampf MP, Gosman GG, Nestler JE, Carson S, Myers EE, Eisenberg E, Legro RS; Eunice Kennedy Shriver National Institute of Child Health and Human Development Cooperative Reproductive Medicine Network. Endometrial shedding effect on conception and live birth in women with polycystic ovary syndrome. Obstet Gynecol. 2012 May;119(5):902-8. doi: 10.1097/AOG.0b013e31824da35c. PMID 22525900
- [Result] Wei D, Shi Y, Li J, Wang Z, Zhang L, Sun Y, Zhou H, Xu Y, Wu C, Liu L, Wu Q, Zhuang L, Du Y, Li W, Zhang H, Legro RS, Chen ZJ. Effect of pretreatment with oral contraceptives and progestins on IVF outcomes in women with polycystic ovary syndrome. Hum Reprod. 2017 Feb;32(2):354-361. doi: 10.1093/humrep/dew325. Epub 2016 Dec 19. PMID 27999118